CLINICAL TRIAL: NCT06578520
Title: Effect of the Use of Dapagliflozin in Diuresis, Natriuresis and in Ultrafiltration and Peritoneal Elimination of Sodium, in Patients With Refractory Heart Failure
Brief Title: Effect of the Use of Dapagliflozin in Patients With Refractory Heart Failure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAPA-DP
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, crossover study, parallel, 2-sequence, 2-period, 2-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): They will receive standard of care plus Dapaglifozin for 8 weeks, after a 4-week wash out, they will receive receive standard of care for another 8 weeks.
  Interventions: Drug: Dapagliflozin
- Group 2 (Experimental): They will receive standard of care for 8 weeks, after a 4-week wash out, they will receive receive standard of care for another 8 weeks plus Dapaglifozin.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg once per day, oral tablets
  Other Names: Forxiga

SUMMARY:
Cross-over, 2-sequence, 2-treatment, 2-period single-centre, phase IV, randomized, open label study.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is a technique that has been successfully used for the treatment of refractory heart failure to diuretics. In patients on PD, the harmful effects of sodium retention become even greater, resulting in fluid overload, hypertension and left ventricular hypertrophy in more than half of the PD population. This is due to the fact that the accumulation of sodium in the skin interstitium would generate an inflammatory environment and, therefore, the activation of growth and fibrogenic factors with a consequent increase in cardiac muscle mass.

In patients with HF receiving PD, therefore, it is necessary to reduce salt intake with diet, as well as to ensure adequate elimination through available medical treatments and elimination of Na through the most appropriate dialysis technique.

In recent years, a new player has joined the treatment of HF: iSGLT2, an oral hypoglycaemic drug. ISGLT2 promotes natriuresis thanks to its well-known mechanism of inhibition of Na and glucose co-transporter. Also promoting excretion of Na at the distal tubule level due to increased tubular osmotic pressure secondary to glycosuria, as well as by direct inhibition of NH3 channels reabsorbing Na and Hydrogens.

The purpose of the study is to analyse whether the use of an SGLT2 inhibitor (Dapagliflozin) in patients with CKD and HF treated with peritoneal dialysis can benefit patients in terms of increased total elimination of sodium and water.

In this study, dapagliflozin will be used together with established drug therapy for patients with HF, including concomitant diuretic therapy.

after randomization, the patient will be divided in two groups and they will receive the study drug or placebo for 8 weeks and, after a 4-week wash out, each patient will switch groups for further 8 weeks to receive standard of care or standard of care plus Dapaglifozin as appropriate.

The study will end with a safety extension study in which all patients will take Dapagliflozin for a further 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Provision of informed consent form prior to any study specific procedures, sampling and analysis.
* Individuals must be ≥ 18 years of age at the time of signing the informed consent
* Individuals must have a confirmed diagnosis of Heart Failure (HF) according to clinical practice guidelines NYHA functional class I-III (with HFrEF or HFpEF).
* In treatment with Peritoneal Dialysis technique
* Chronic Kidney Disease (eGFR < 60 ml/min/m2 CKD-EPI formula)
* PD vintage of more than 30 days
* On stable doses of furosemide, or alternative loop diuretic for 14 days
* On stable HF therapy for at least 1 month prior to consent
* No hospitalizations for HF for at least 1 month prior to consent

Exclusion Criteria:

* Limited life expectancy (less than 1 year) based on investigator's clinical judgement.
* Patients without indication of beginning treatment with Dapagliflozin according to the Data Sheets and Consumer Medicine Information.
* Malignancy (with active treatment) or other life-threatening disease
* Patients in whom proper study compliance cannot be guaranteed
* Rejection or revocation of informed consent
* Current acute decompensated HF, hospitalization due to decompensated HF, myocardial infarction, unstable angina, stroke or transient ischemic attack within 1 month prior to enrollment.
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting or valvular repair/replacement) within 1 month prior to enrollment or planned to undergo any of these operations after randomization.
* Implantation of a Cardiac Resynchronization Therapy (CRT) device or Implantable Cardioverter Defibrillator (ICD) within 1 month prior to enrollment or intent to perform atrial fibrillation ablation or to implant a CRT or ICD device.
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or transplantation or implantation expected after randomization
* Pregnant or breast-feeding women
* Type 1 Diabetes
* Residual urine volume less than 500ml daily or reduction in urinary output by 24 hours (< 30% compared to previous routine control) within 30 days prior to consent
* Patients with amputated limbs will be excluded of bioimpedance analysis.
* Participation in another clinical study with an investigational product during the last 3 months.
* Patients with a known hypersensitivity to Dapagliflozin or any of the excipients of the product.
* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference of the sum between 24-h natriuresis and the daily sodium elimination in the peritoneal effluent (mEq/L) in the 3rd (8th week) visit control compared with the 6th (20th week)visit control. | Through study completion, an average of 4 months
  To explore the effect of iSGLT2 in natriuresis and the peritoneal elimination of sodium in patients with CKD and refractory HF treated with peritoneal dialysis.

SECONDARY OUTCOMES:
Mean difference of the sum between the volume of diuresis in 24 hours and the daily peritoneal effluent ultrafiltration rate (ml/24hours) in the 3rd (8th week) visit control compared with the 6th (20th week) visit control. | Through study completion, an average of 4 months
  To explore the effect of the use of iSGLT2 in diuresis and, in the peritoneal net ultrafiltration in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean difference of the sum between the volume of diuresis in 24 hours and the daily peritoneal effluent ultrafiltration rate (ml/24hours) in the 2nd (4th week) visit control compared with the 5th (16th week) visit control. | Through study completion, an average of 4 months
  To explore the effect of the use of iSGLT2 in diuresis and, in the peritoneal net ultrafiltration in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean difference of the sum between 24-h natriuresis and the daily sodium elimination in the peritoneal effluent (mEq/L) in the 2nd visit control compared with the 5th visit control. | Through study completion, an average of 4 months
  To explore the effect of iSGLT2 in natriuresis and the peritoneal elimination of sodium in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean difference between the hydration percentage: Total Body Water%, Extracellular Water% , Intracellular Water%, Plasma Fluid, Interstitial Fluid by bioimpedance in the 3rd visit control compared with the 6th visit control. | Through study completion, an average of 4 months
  To explore the effect of the use of iSGLT2 in the normalization of extracellular volume in patients with CKD and refractory HF treated with peritoneal dialysis.
Collection of chemistry parameters: Mean change and standard deviations in Peritoneal Fluid Glucose Ratio and Sodium concentration in the effluent peritoneal dialysis fluid sample in the 3rd visit control compared with the 6th visit control. | Through study completion, an average of 4 months
  To evaluate the effect of the use of iSGLT2 in Glucose and sodium homeostasis in the peritoneal fluid effluent in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean change and standard deviations in Peritoneal Fluid Glucose Ratio (D4/D0) and Sodium (mEq/24hr) concentration in the effluent peritoneal dialysis fluid sample in the 2nd visit control compared with the 5th visit control. | Through study completion, an average of 4 months
  To evaluate the effect of the use of iSGLT2 in Glucose and sodium homeostasis in the peritoneal fluid effluent in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean Difference in NYHA Classification, Ultrasounds parameters for the evaluation of venous congestion and BNP (ng/ml), CA 125 (ng/ml) in the blood sample in the 3rd visit control compared with the 6th visit control. | Through study completion, an average of 4 months
  To evaluate the effect of the use of iSGLT2 in the clinical and laboratory parameters in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean difference in Ca125 (U/min), IL-6 (pg/min), in the effluent peritoneal dialysis fluid sample in the 3rd visit control compared with the 6th visit control. | Through study completion, an average of 4 months
  To study the effect of the use of iSGLT2 in the inflammatory state of the peritoneal membrane in patients with CKD and refractory HF treated with peritoneal dialysis.
Mean Change in the total amount of loop diuretic and thiazide treatment (mg/daily) in the 3rd visit control compared with the 6th visit control. | Through study completion, an average of 4 months
  To evaluate the effect of the use of iSGLT2 in dose reduction of diuretics and the need for diuretic therapy in patients with CKD and refractory HF treated with peritoneal dialysis.

OTHER OUTCOMES:
Collection of serious adverse events. The proportion of patients treated with DAPA presenting these adverse events, in comparison to the patients non-treated with DAPA, at the visit control 3rd, 6th and 8th. | Through study completion, an average of 4 months
  To explore the safety of iSGLT2 in patients with CKD and refractory HF treated with peritoneal dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montomoli, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No